CLINICAL TRIAL: NCT06026995
Title: Clinical Study on the Effectiveness and Safety of PEG-rhG-CSF in Mobilizing Autologous Hematopoietic Stem Cells for Lymphoma and Multiple Myeloma
Brief Title: Clinical Study on PEG-rhG-CSF in Mobilizing Autologous Hematopoietic Stem Cells
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yao Liu, Director, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-PBSCT-02
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: PEG-rhG-CSF
- control group (Active Comparator)
  Interventions: Drug: RhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — Subcutaneous injection with a fixed dose of 12 mg
  Arms: experimental group
Drug: RhG-CSF — Inject rhG-CSF 5-10 μg/kg subcutaneously every day
  Arms: control group

SUMMARY:
This study is a randomized controlled, open and multi-center clinical study. Patients who meet the selection criteria and do not meet the exclusion criteria are randomly given PEG-rhG-CSF with a fixed dose of 12mg when white blood cells reach the lowest point, or given rhG-CSF with a daily mobilization of 5-10μ g/kg until the collection is completed, so as to evaluate the effectiveness and safety of PEG-rhG-CSF in mobilizing autologous stem cells for lymphoma and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old, regardless of sex;
2. Patients with lymphoma and multiple myeloma who need autologous hematopoietic stem cell transplantation;
3. KPS score ≥70;
4. creatinine clearance rate ≥ 50mL/min, total bilirubin level < 1.5mg/dL, ALT and AST < 2 times the upper limit of normal value;
5. Absolute neutrophil count (ANC)≥1.5×109/L, platelet count ≥80×109/L, Hb≥ 75g/L, WBC ≥ 3.0× 109/L;
6. Patients can tolerate chemotherapy;
7. No active infection before chemotherapy;
8. The patient voluntarily participated in this trial and signed the informed consent form;
9. The researcher thinks that the subjects can benefit.

Exclusion Criteria:

1. Those who have previously received allogeneic or autologous hematopoietic stem cell transplantation;
2. Serious or uncontrolled virus infection: HIV, syphilis positive;
3. Severe dysfunction of internal organs;
4. severe mental or nervous system diseases;
5. allergic to PEG-rhG-CSF, rhG-CSF and other preparations or proteins expressed in Escherichia coli;
6. pregnant or lactating female patients; Women of childbearing age refuse to accept contraceptive measures; Those who plan to become pregnant during the study period;
7. The researcher judges other subjects who are not suitable to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with CD34+ cells ≥2×106/kg | 28 days
  The proportion of patients with CD34+ cells ≥2×106/kg

SECONDARY OUTCOMES:
CD34+cell count | 28 days
  CD34+cell count
Acquisition times | 28 days
  The number of times a patient needs to collect a sufficient number of CD34+ cells
Mobilization time | 28 days
  Time interval from mobilization to collection
Hematopoietic reconstruction time after transplantation | 3 months
  Hematopoietic reconstruction time after transplantation
complication | 3 months
  complication

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No